CLINICAL TRIAL: NCT01009710
Title: Preoperative Cerebrospinal Fluid (CSF) Levels of Hypocretin and Recovery After Hip Surgery With Combined Spinal and General Anesthesia
Brief Title: Measured Hypocretin Levels and Recovery After Hip Surgery
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Anthony Doufas, MD, PhD, Stanford University
Other Study IDs: SU-07162009-3301; 16339
Record Dates: First submitted 2009-11-05; First posted 2009-11-09 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Osteoarthritis, Hip
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
A specific group of neurons in the brain produces hypocretin, a peptide which has been established as an important regulator of sleep and wakefulness. Activation of these neurons (increased hypocretin) stabilizes wakefulness; impairing or blocking these neurons (decreased hypocretin) promotes sleep. Evidence suggests that these neurons may be involved in the hypnotic properties of several anesthetics, and play a role in the induction and emergence from anesthesia. In humans there is a considerable inter-individual variability in hypocretin levels. This study aims to investigate how hypocretin levels affect the anesthetic care and recovery of patients undergoing elective hip surgery.

ELIGIBILITY:
Inclusion Criteria:- Adult (18 years of age or older)

* Male or female
* Scheduled for elective total hip arthroplasty at the Stanford Orthopedic Clinic.
* Comprehend spoken and written English Exclusion Criteria:- ASA physical status > III (patients with severe systemic disease)
* Diagnosed psychiatric disease (except mild depression)
* Any diagnoses CNS disease or dementia
* History of stroke
* History of untreated thyroid disease
* Difficulty in airway management (ventilation and/or intubation)
* Body Mass Index (BMI) > 35 kg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective total hip arthroplasty through the Stanford Orthopedic Clinic.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2009-07; Primary Completion 2013-12 (Actual); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Anesthetic Recovery Times | 0-72 hours after surgery
  recovery from anesthesia will be measured by short-term outcomes like time to tracheal extubation and response to verbal commands, as well as by psycho-vigilance testing up to 72 hours postoperatively

SECONDARY OUTCOMES:
sensitivity to sevoflurane during inhalation induction to anesthesia, determined by bispectral index of the EEG | during anesthetic induction
  pharmacodynamic analysis of bispectral index of the EEG response to sevoflurane
pain and sleepiness | from 0-72 hours after surgery
  assessment of pain and sleepiness using the numerical rating scale (0-10) during the 72 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Doufas, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States